CLINICAL TRIAL: NCT06530836
Title: Chronic Diarrhea Owing to Underlying Microscopic Colitis: Diagnosis Challenges and Size of the Problem
Brief Title: Chronic Diarrhea Owing to Underlying Microscopic Colitis
Status: Active, not recruiting | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ayman Magd Eldin Mohammad Sadek, Associate Professor of Internal Medicine, Zagazig University
Other Study IDs: ZU-IRB#239/17-March-2024
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Chronic Diarrhea; Microscopic Colitis
MeSH Terms: conditions — Colitis, Microscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to search for accurate diagnoses for patients with chronic diarrhea and assess the prevalence of microscopic colitis. The main question[s] it aims to answer [is/are]:

Does microscopic colitis account for a significant portion of patients with chronic diarrhea?

Participants will subjected to:

* Routine laboratory examination.
* Colonoscopy: A total colonoscopy will be done with visualization of the terminal ileum. Biopsies will be taken from each segment of the colon and any abnormal appearing areas, the right-sided colon (cecum, ascending colon, and transverse colon), the left-sided colon (descending colon and sigmoid colon), and the rectum.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic watery diarrhea

Exclusion Criteria:

* Infectious colitis.
* Inflammatory bowel diseases (ulcerative colitis, Crohn's disease, and indeterminate colitis).
* Systemic disease associated with chronic diarrhea, e.g. Diabetes mellitus and Thyroid disease.
* Drugs causing chronic diarrhea, e.g. antibiotics, antidepressants, and angiotensin-converting enzyme inhibitors.
* Chronic diarrhea of decreased digestion as in pancreatic insufficiency and bile acid deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presented with chronic diarrhea in the outpatient clinic or the inward in the Gastroenterology and Hepatology unit in the Internal Medicine Department, Zagazig University hospitals from January 2024 to January 2025
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Chronic Diarrhea Diagnosed with Microscopic Colitis | 6 weeks
  Diagnostic criteria for the diagnosis of microscopic colitis include increased chronic inflammatory infiltration in the lamina propria, increased intraepithelial lymphocytes (IELs), degeneration of surface epithelium, and increased mitosis in crypts.

SECONDARY OUTCOMES:
Rate of Lymphocytic and Collagenous Types of Microscopic Colitis in Individuals Experiencing Chronic Diarrhea | 2 weeks
  Over 20 IELs per 100 inter-cryptal epithelial cells (normal <1-5/100) were required for the diagnosis of lymphocytic colitis.
  For collagenous colitis, subepithelial collagen band thickness was measured by ocular micrometer in specimens stained with Masson's Trichrome. Specimen thickness over 10 μm was required for the diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Sadek, MD, Study Director — Associate Professor of Internal Medicine - Zagazig University
Locations (1):
- Zagazig University Hospital, Zagazig, Sharqia Province, Egypt